CLINICAL TRIAL: NCT07143149
Title: Effect of the Intelligent Lipid Management Decision-support System on 1-year LDL-C Target Achievement in Ischemic Stroke or TIA Patients Under Evolocumab Treatment in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2025-210 -02
Record Dates: First submitted 2025-08-04; First posted 2025-08-27 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack (TIA)
Keywords: ischemic stroke; LDL-C; LDL-C Target Achievement; the Intelligent Lipid Management Decision-support System; Evolocumab
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Intelligent Lipid Management Decision-support System (Experimental): Doctor's Side: Long-term lipid management support based on guidelines/consensus• Provides lipid management pathways based on guidelines/consensus to ensure clinical decisions align with the latest standards.• Combines individualized patient data to offer intelligent lipid management and medication suggestions.• Provides medical education support to enhance doctors' awareness of guidelines, consensus, and management strategies.Patient's Side: Personalized lipid risk assessment and regular reminders• Based on the lipid test reports uploaded by patients via photos, provides lipid test reports tailored to the patient's risk stratification.• Uses digital tools to regularly remind patients, optimizing follow-up adherence and medication compliance.
  Interventions: Device: the Intelligent Lipid Management Decision-support System
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Device: the Intelligent Lipid Management Decision-support System — Doctor's Side: Long-term lipid management support based on guidelines/consensus• Provides lipid management pathways based on guidelines/consensus to ensure clinical decisions align with the latest standards.• Combines individualized patient data to offer intelligent lipid management and medication suggestions.• Provides medical education support to enhance doctors' awareness of guidelines, consensus, and management strategies.Patient's Side: Personalized lipid risk assessment and regular reminders• Based on the lipid test reports uploaded by patients via photos, provides lipid test reports tailored to the patient's risk stratification.• Uses digital tools to regularly remind patients, optimizing follow-up adherence and medication compliance.
  Arms: the Intelligent Lipid Management Decision-support System

SUMMARY:
This study will conduct a cluster randomized controlled trial to Evaluate whether the Intelligent Lipid Management Decision-support System can increase the proportion of patients 1-year target achievement (<1.8 mmol/L) in acute ischemic stroke or TIA patients under Evolocumab treatment within 12 months post-intervention.

DETAILED DESCRIPTION:
Large scale randomized trials and systematic reviews have established the efficacy of lipid lowering therapy for acute ischemic stroke. However, adherence to these evidence-based performance measures is suboptimal and gaps in adherence to guideline recommended care are even greater in China. Multifaceted quality improvement interventions that address the barriers to care are effective in changing physician practices. Quality improvement interventions have demonstrated that stroke care quality can be improved by conducting interventions such as using clinical pathways, training physicians on evidence-based guidelines, auditing care delivery, and providing timely feedback.

Aim: To Evaluate whether the Intelligent Lipid Management Decision-support System can increase the proportion of patients 1-year target achievement (<1.8 mmol/L) in acute ischemic stroke or TIA patients under Evolocumab treatment within 12 months post-intervention.

Intervention: The Intelligent Lipid Management Decision-support System primarily consists of an evidence-based clinical pathway. The evidence-based clinical pathway was written by a panel of stroke experts according to the published statements in peer-reviewed literature, consensus statements and guidelines. It was integrated into the care plan of each eligible stroke admission.

Eligible hospitals in china, stratified by economic-geographical regions, will be randomized into either the intervention group or the control group.

ELIGIBILITY:
Inclusion Criteria

1. Age≥18 years as of the screening date;
2. Patients with non-cardioembolic ischemic stroke or TIA within 3 months prior to the screening date;
3. Prescribed Evolocumab at physician's discretion;
4. Signed informed consent.

Exclusion Criteria:

1. Intracranial hemorrhagic diseases: such as cerebral hemorrhage, subarachnoid hemorrhage, etc.;
2. Patients confirmed by baseline head CT or MRI to have hemorrhage or other pathological brain diseases, such as vascular malformations, tumors, abscesses, or other common non-ischemic brain diseases (such as multiple sclerosis);
3. Silent cerebral infarction without signs and symptoms;
4. Participation in a clinical trial of another drug or device in the past 3 months or ongoing at the time of the screening date;
5. Any prior use of Evolocumab or other PCSK9 inhibitor treatments within the past 6 months prior to the screening date;
6. Life expectancy <12 months or unable to complete the research for other reasons as of the screening date;
7. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders;
8. Refusal to participate in the enrollment survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of acute ischemic stroke or TIA patients achieving LDL-C <1.8 mmol/L at 1 year with Evolocumab treatment | at 365 days (±14days）
  To Evaluate whether the Intelligent Lipid Management Decision-support System can increase the proportion of patients 1-year target achievement (<1.8 mmol/L) in acute ischemic stroke or TIA patients under Evolocumab treatment within 12 months post.

SECONDARY OUTCOMES:
Percentage decrease from baseline in LDL-C at each visit (3 months and 12 months). | at 90 days (±7 days) and 365 days (±14 days）
  To investigate the LDL-C percentage decrease from baseline in patients with ischemic stroke or TIA using Evolocumab at 3 months and 12 months.
Duration (in months) of maintaining LDL-C levels within the target range (<1.8 mmol/L) within 12 months post-intervention. | at 365 days (±14 days）
  Duration (in months) of maintaining LDL-C levels within the target range (<1.8 mmol/L) among patients receiving Evolocumab treatment, within 12 months post-intervention.
Proportion of acute ischemic stroke or TIA patients achieving LDL-C <1.8 mmol/L at 3 months with Evolocumab treatment | at 90 days（±7 days）
  To investigate whether the Intelligent Lipid Management Decision-support System can increase the proportion of patients achieving target LDL-C levels at 3 months under Evolocumab treatment with ischemic stroke or TIA in China
Frequency of subcutaneous Evolocumab injections at 3-month follow-up | at 90 days （±7 days）
  Frequency of subcutaneous Evolocumab injections at 3-month follow-up as a measure of treatment persistence in ischemic stroke/TIA patients
Incidence rate of stroke recurrence and cardiovascular outcome events | at 90 days (±7 days) and 365 days (± 14 days)
  Stroke recurrence and cardiovascular outcome events at each visit (3 months and 12 months) following the administration of Evolocumab in patients with ischemic stroke or TIA.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No